CLINICAL TRIAL: NCT04021407
Title: Laryngeal Mask Airway Versus Air Q Laryngeal Airway in Dacryocystorhinostomy
Brief Title: Laryngeal Mask Airway Versus Air Q Laryngeal Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, ashraf magdy eskandr, assistant professor of anesthesia, icu, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: LMA versus Air Q
Record Dates: First submitted 2019-07-10; First posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Airway Devices
Keywords: AirQ; LMA; dacrocystorhinostomy surgery

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: Participiant Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LMA (Active Comparator): 36 patients were ventilated with LMA during dacryocystorhinostomy surgery
  Interventions: Device: LMA group
- AirQ (Active Comparator): 36 patients each were ventilated with air Q airway during dacryocystorhinostomy surgery
  Interventions: Device: AirQ group

INTERVENTIONS:
Device: LMA group — patients were ventilated with LMA
  Arms: LMA
Device: AirQ group — patients were ventilated with AirQ airway
  Arms: AirQ

SUMMARY:
Nowadays, supraglottic airway devices are simple and effective alternatives to endotracheal intubation. Both laryngeal mask airway LMA and air-Q airway are supraglottic airway devices that can be used to maintain and protect airways from aspiration of secretions and blood during DCR surgery. The present study was designed to compare standard LMA versus air Q as regards the sealing effect and aspiration of blood in DCR surgery.

DETAILED DESCRIPTION:
72 patients were divided into two groups, 36 patients each, named LMA group, and air Q group according to supraglottic devices used. The following parameters were recorded in both studied groups, continuous Electrocardiography (ECG), heart rate (HR), means arterial pressure (MAP), arterial oxygen saturation (SpO2), end tidal carbon di-oxide (PCO2)..Oro pharyngeal leak pressure in (cmH2O), exhaled tidal volume in (ml), leak volume in (ml), leak fraction in (%) number of shifting from LMA to air Q or ETT and shifting from air Q to LMA or ETT was recorded with absence or presence of surgical blood on The undersurface of the device used.

ELIGIBILITY:
Inclusion Criteria:

* Both sex
* Age: 18-60 years
* ASA I-II
* Patients scheduled for dacryocystorhinostomy surgery

Exclusion Criteria:

* Any pathology of the neck, upper respiratory tract, upper alimentary tract
* Patients with a history of gastric regurgitation, heartburn
* Morbid obese,
* Patients with esophageal reflux (hiatus hernia)
* Anticipating difficult airway management
* Patients with coagulation disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Oro pharyngeal leak pressure in (cmH2O) | Just after insertion of supraglottic airway devices
  By setting the pop-off valve to limit peak airway pressure to 40 cm H2O and allowing airway pressure to increase at a fresh gas flow of 3 L/min until audible noise was heard over the mouth and no further increase in airway pressure is observed.

SECONDARY OUTCOMES:
Leak fraction in (%) | Just after insertion of supraglottic airway devices
  Leak fraction in (%)( Leak was calculated by subtracting the expiratory volume from the inspiratory volume and expressed as a fraction of the inspiratory volume). were evaluated just before surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Ashraf Eskandr, Shibīn al Kawm, Monufia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No